CLINICAL TRIAL: NCT00001085
Title: A Randomized, Double-Blind, Phase II Study of 141W94 (VX-478) Monotherapy vs. 141W94 (VX-478) Plus ZDV Plus 3TC in HIV Infected Individuals
Brief Title: A Study of 141W94 Used Alone or in Combination With Zidovudine Plus 3TC in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 347; 11317 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; HIV Protease Inhibitors; Lamivudine; RNA, Viral; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — amprenavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Amprenavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To determine the proportion of patients whose plasma HIV-1 RNA level remains below a detectable level (less than 500/ml) after 24 weeks of study therapy with either 141W94 monotherapy or 141W94 plus zidovudine (ZDV) and lamivudine (3TC). To determine the safety and tolerability of 141W94 monotherapy and the combination of 141W94 plus 3TC in patients with HIV infection.

Although dramatic inhibition of HIV-1 replication is achieved with ritonavir or indinavir monotherapy, in both cases maximum suppression required combination treatment together with nucleoside analog RT inhibitors. This study tests the hypothesis that monotherapy with 141W94 doses that result in Cmin levels far in excess of the IC90 corrected for plasma protein binding for HIV-1 can achieve the same virologic and immunologic effects in terms of magnitude and durability, as has been observed with combinations of other protease inhibitors plus nucleoside analogs.

DETAILED DESCRIPTION:
Although dramatic inhibition of HIV-1 replication is achieved with ritonavir or indinavir monotherapy, in both cases maximum suppression required combination treatment together with nucleoside analog RT inhibitors. This study tests the hypothesis that monotherapy with 141W94 doses that result in Cmin levels far in excess of the IC90 corrected for plasma protein binding for HIV-1 can achieve the same virologic and immunologic effects in terms of magnitude and durability, as has been observed with combinations of other protease inhibitors plus nucleoside analogs.

In this randomized, double-blind study, patients' HIV RNA is screened 30 days prior to entry. Patients satisfying enrollment criteria must have been on a stable antiretroviral regimen for 30 days prior to study screening and remain on the same regimen until entry. Patients are stratified based on the screening HIV-1 RNA copy number obtained within 30 days of entry: 5,000 - 50,000 copies/ml versus greater than 50,000 copies/ml. In addition, patients are stratified based on previous antiretroviral use: naive versus experienced. Patients are randomized to one of 2 treatment arms: Arm A - 141W94, plus Zidovudine (ZDV) and Lamivudine (3TC) or Arm B - 141W94, plus ZDV placebo and 3TC placebo.

[AS PER AMENDMENT 8/25/97: Patients assigned to the monotherapy arm are advised to discontinue their study medication immediately and initiate antiretroviral therapy with indinavir, nevirapine, stavudine and 3TC, as outlined in ACTG 347 roll-over protocol, ACTG 373. Patients in the three-drug arm continue on study therapy.] [AS PER AMENDMENT 12/19/97: Patients receive study treatment for 56 weeks and are followed through week 68.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia is required for all patients who have a CD4 cell count <= 200 cells/mm3.
* Topical and/or oral antifungal agents, except for those listed in excluded medications.
* Treatment, maintenance or chemoprophylaxis with approved agents for opportunistic infections as clinically indicated, unless listed in excluded medications.
* All antibiotics as clinically indicated.
* Systemic corticosteroid use for <= 21 days for acute problems is permitted as medically indicated; chronic systemic corticosteroid use is not permitted.
* Recombinant erythropoietin and granulocyte colony-stimulating factor as medically indicated.

Regularly prescribed medications such as:

* antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives (a barrier method is also required for this study), megestrol acetate, testosterone or any other medications, as medically indicated.
* Alternative therapies such as vitamins, acupuncture and visualization techniques are permitted (excluding herbal medications).

NOTE:

* Patients should report the use of these therapies; alternative therapies will be recorded.

Patients must have:

* HIV-1 infection as documented by ELISA and confirmed.
* >= 5,000 HIV-1 RNA copies/ml (within 30 days prior to study entry).
* CD4 cell count >= 50 cells/mm3 within 60 days prior to study entry.
* Signed, informed consent for patients < 18 years of age.

Prior Medication: Required:

* Patients must be on a stable antiretroviral regimen for 30 days prior to study screening and remain on the same regimen until entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Any active infection requiring acute treatment within 14 days prior to entry.
* A malignancy that requires systemic therapy other than minimal Kaposi's sarcoma.

NOTE:

* Patients with minimal Kaposi's sarcoma, defined as <= 5 cutaneous lesions and no visceral disease or tumor-associated edema, will be allowed to enroll as long as they do not require systemic therapy for Kaposi's sarcoma.

Patients with the following prior symptoms and conditions are excluded:

* Inability to tolerate ZDV 500-600 mg daily if ZDV was administered previously. Intolerance to ZDV is defined as any grade toxicity that resulted in a dose reduction or termination of ZDV.

Prior Medication:

Excluded:

* Any 3TC therapy prior to entry.
* Any HIV-1 protease inhibitor therapy prior to study entry (e.g., saquinavir, ritonavir, indinavir, nelfinavir, 141W94).
* Any immunomodulator therapy within 30 days prior to entry.
* Active immunization within 30 days prior to entry.
* Any antiretroviral therapy change within 30 days prior to study screening.

  1. Concurrent use of non-protocol specified antiretroviral agents; either investigational or licensed.
* Immunomodulators that affect immunologic or virologic indices such as systemic corticosteroids, thalidomide, or cytokines.
* Concomitant use of rifabutin and/or rifampin.
* Investigational drugs other than 141W94/VX-478.
* Systemic cytotoxic chemotherapy.
* Oral astemizole (Hismanal), carbamazepine (Tegretol), dexamethasone (Decadron), ketoconazole (Nizoral), itraconazole (Sporanox), phenobarbital, phenytoin (Dilantin), terfenadine (Seldane), cisapride (Propulsid), triazolam (Halcion) and midazolam (Versed).
* Herbal medications.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94
Dates: Study Completion 1998-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murphy R, Study Chair; Gulick R, Study Chair
Locations (15):
- United States (15):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Murphy RL, Gulick RM, DeGruttola V, D'Aquila RT, Eron JJ, Sommadossi JP, Currier JS, Smeaton L, Frank I, Caliendo AM, Gerber JG, Tung R, Kuritzkes DR. Treatment with amprenavir alone or amprenavir with zidovudine and lamivudine in adults with human immunodeficiency virus infection. AIDS Clinical Trials Group 347 Study Team. J Infect Dis. 1999 Apr;179(4):808-16. doi: 10.1086/314668. PMID 10068575
- [Background] Murphy R, Degruttola V, Gulick R, D'Aquila R, Eron J, Sommadossi JP, Smeaton L, Currier J, Tung R, Kuritzkes D. 141W94 with or without zidovudine/3TC in patients with no prior protease inhibitor or 3TC therapy-ACTG 347. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:175 (abstract no 512)
- [Background] Eron JJ Jr, Smeaton LM, Fiscus SA, Gulick RM, Currier JS, Lennox JL, D'Aquila RT, Rogers MD, Tung R, Murphy RL. The effects of protease inhibitor therapy on human immunodeficiency virus type 1 levels in semen (AIDS clinical trials group protocol 850). J Infect Dis. 2000 May;181(5):1622-8. doi: 10.1086/315447. Epub 2000 Apr 26. PMID 10783117
- [Background] Eron J, Smeaton L, Degruttola V, Schock J, Fiscus S, Tung R, Gulick R, Murphy R. The effects of amprenavir (APV) alone or in combination with ZDV/3TC, on HIV-1 levels in semen: a substudy of ACTG 347. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:109 (abstract no 222)